CLINICAL TRIAL: NCT05460078
Title: An Evaluation of Virtual Psychiatric Transition of Care Offered in Behavioral Health Settings
Brief Title: An Evaluation of Virtual Psychiatric Transition of Care Offered in Behavioral Health
Acronym: VPTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00082500
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-05

CONDITIONS: Mental Health Issue
Keywords: behavioral health symptoms

STUDY DESIGN:
Intervention Model Description: stepped-wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual program (Experimental): Seen at a location where the virtual program is being offered
  Interventions: Behavioral: Virtual Psychiatric Transition of Care Program
- Standard care (No Intervention): Seen at a location where standard care is offered

INTERVENTIONS:
Behavioral: Virtual Psychiatric Transition of Care Program — Behavioral Health facility or units that have discharged patients meeting inclusion criteria will be randomly assigned as either an intervention or standard care site. Intervention sites will be those using the VPTC program. This evaluation design will integrate into current workflows for the measurement of outcomes. Prior to discharge, patients may be referred to the VPTC program if they report residency or shelter in North Carolina, are 18 years of age or older on the day of discharge and can access virtual care (phone/video).
  The VPTC program is defined by:
  * Psychiatric consultation
  * Medication management services with pharmacological consultation
  * following of Health Coaching participation and provide treatment recommendations
  * Tracking of behavioral health symptoms and provide treatment recommendations
  * Health coaching; Psychoeducational support
  * Treatment and safety planning
  * Assistance connecting with an outpatient care provider
  Arms: Virtual program

SUMMARY:
The primary objective is to evaluate the effectiveness of a post inpatient discharge virtual psychiatric care team compared to standard care, to reduce 30-day all cause non-elective acute care utilization (Emergency Department (ED), observation, and inpatient encounters).

DETAILED DESCRIPTION:
The foundational idea for the Virtual Psychiatric Transition of Care (VPTC) program came from the Atrium Health Hospital at Home care model which has garnered wide acclaim and financial support in the acute care world. A behavioral health care team comprised of licensed clinicians (Behavioral Health Professionals), health coaches, a consulting psychiatric pharmacist and psychiatric providers follow patients for 45 days or more depending on patient need after their acute care encounter. Patient enrolled in the VPTC program will receive the following core components: Introduction to the patient follow-up process, psychosocial assessment, tracking and treatment recommendations for (residential movement, nutrition, sleep hygiene, stress management, pain management, perinatal/postpartum mood disorders, substance abuse), tracking and treatment recommendations for behavioral health symptoms (depression, anxiety, suicidal ideation, etc.), placement into an appropriate case management program if needed, navigation to additional psychiatric or substance use services if needed, and motivational interviewing and brief therapeutic recommendations if needed.

For patients that have attempted suicide, they will begin the VPTC program following the zero suicide pathway. The Atrium Health Behavioral Health Service Line created the 'Zero Suicide pathway', in 2019 for those patients identified as "high risk" for suicide when leaving inpatient units. Zero Suicide is a national movement sponsored by the 2012 National Strategy for Suicide Prevention, National Alliance for Suicide Prevention, Suicide Prevention Resource Center and the Substance Abuse and Mental Health Services Administration (SAMHSA). It is a programmatic approach to keep patients from falling through the cracks in a fragmented and disconnected healthcare system and is based on the belief that suicide is preventable, and suicide deaths are not fated. Since access to mental health services is constrained in our community, patients often fall through the cracks when transitioning between points of care.

ELIGIBILITY:
Inclusion Criteria:

* Residency or shelter in North Carolina
* 18 years of age or older on the day of discharge
* Access virtual care (phone/video)
* Discharged from a behavioral health hospital or a behavioral health unit

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7526 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Roberge, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - Atrium Health Behavioral Health Davidson - Mountain Laurel, Charlotte, North Carolina
  - Atrium Health Behavioral Health Davidson - River Birch, Charlotte, North Carolina
  - Carolinas Medical Center Main - 6B, Charlotte, North Carolina
  - Atrium Health Behavioral Health Charlotte - ED Obs, Charlotte, North Carolina
  - Atrium Health Behavioral Health Charlotte - North and South, Charlotte, North Carolina
  - Atrium Health Behavioral Health Davidson - Frasier Fur, Davidson, North Carolina
  - Atrium Health Kings Mountain Psychiatry, Kings Mountain, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Program: Seen at a location where the virtual program is being offered
  Virtual Psychiatric Transition of Care Program: Behavioral Health facility or units that have discharged patients meeting inclusion criteria will be randomly assigned as either an intervention or standard care site. Intervention sites will be those using the VPTC program. This evaluation design will integrate into current workflows for the measurement of outcomes. Prior to discharge, patients may be referred to the VPTC program if they report residency or shelter in North Carolina, are 18 years of age or older on the day of discharge and can access virtual care (phone/video).
  The VPTC program is defined by:
  * Psychiatric consultation
  * Medication management services with pharmacological consultation
  * following of Health Coaching participation and provide treatment recommendations
  * Tracking of behavioral health symptoms and provide treatment recommendations
  * Health coaching; Psychoeducational support
  * Treatment and safety planning
  * Assistance connecting with an outpatient care provider
Period: Overall Study
Arm/Group | Virtual Program | Standard Care
Started (Discharges identified as eligible) | 3616 | 3910
Completed (Actually enrolled in the program) | 1382 | 3910
Not Completed | 2234 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Program | Standard Care | Total
Number analyzed (Participants) | 3616 | 3910 | 7526
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (13.6) | 37.3 (14.5) | 37.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1546 | 2011 | 3557
  Male | 2070 | 1899 | 3969
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 1557 | 1620 | 3177
  American indian | 38 | 37 | 75
  Asian | 63 | 60 | 123
  Caucasian | 1786 | 1970 | 3756
  Multi-Race | 68 | 93 | 161
  Other | 7 | 10 | 17
  Unknown | 97 | 120 | 217
Region of Enrollment [Number; unit: participants]
  United States | 3616 | 3910 | 7526

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All Cause Non-elective Acute Care Post Discharge Utilization Within 30 Days
Description: 30-day all cause non-elective acute care post discharge utilization (Emergency Department (ED), inpatient, and observation encounters)
Time Frame: day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Program | Standard Care
Number analyzed (Participants) | 3616 | 3910
Participants | 941 | 973
Statistical Analysis 1: Comparison: Virtual Program vs Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.16 to 1.68]

2. Secondary Outcome: 60-day All Cause Non-elective Acute Care Utilization
Description: 60-day all cause non-elective acute care utilization (ED visits, observation, and inpatient encounters)
Time Frame: day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Program | Standard Care
Number analyzed (Participants) | 3616 | 3910
Participants | 1257 | 1270
Statistical Analysis 1: Comparison: Virtual Program vs Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.18 to 1.65]

3. Secondary Outcome: 45-day Behavioral Health Acute Care Utilization
Description: 45-day behavioral health acute care utilization (BH unit or BH ED)
Time Frame: day 45
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Program | Standard Care
Number analyzed (Participants) | 3616 | 3910
Participants | 556 | 622
Statistical Analysis 1: Comparison: Virtual Program vs Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.54 to 2.48]

4. Secondary Outcome: 45-day All Cause Non-elective Acute Care Utilization
Description: 45-day behavioral health acute care utilization (ED visits, observation, and inpatient encounters)
Time Frame: day 45
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Program | Standard Care
Number analyzed (Participants) | 3616 | 3910
Participants | 1124 | 1138
Statistical Analysis 1: Comparison: Virtual Program vs Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.17 to 1.66]

ADVERSE EVENTS:
Time Frame: up to 23 Months
Arm/Group | Virtual Program | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/3616 | 0/3910
Serious Adverse Events (participants affected / at risk) | 0/3616 | 0/3910
Other Adverse Events (participants affected / at risk) | 0/3616 | 0/3910

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05460078/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT05460078/ICF_001.pdf